CLINICAL TRIAL: NCT06235008
Title: PAthwAy of Dyspneic patIent in Emergency in the North-east Region
Brief Title: PAthwAy of Dyspneic patIent in Emergency in the North-east Region (North-East PArADIsE)
Acronym: N_E_PARADISE
Status: Not yet recruiting | Type: Observational
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Clinical Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2020PI059
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational retrospective multi-center study in patients managed for acute dyspnea by Emergency department medical team.

The main aim of the study is to evaluate factors associated with mortality risks in patients managed for acute dyspnea by an Emergency department medical team, overall, as well as in subgroups of interest (male/female, age categories, mode of admission and comorbidities).

ELIGIBILITY:
Inclusion Criteria:

* Man or women ≥ 18 years
* Patients with acute dyspnea cared by a medical team of the emergencies of CHRU of Nancy, CHR Metz-Thionville and CH d'Epinal.

Exclusion Criteria:

* Cardiorespiratory arrest before medical management by the Emergency Department team
* Adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute dyspnea cared by a medical team of the emergencies of CHRU of Nancy, CHR Metz-Thionville and CH d'Epinal
Sampling Method: Non-Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Within 5 years following hospital discharge

SECONDARY OUTCOMES:
Main diagnosis during the initial hospitalization | Within hospital stay, maximum 21 days
Mismatch between diagnosis in the Emergency department and at discharge | Within hospital stay, maximum 21 days
  Difference between the diagnosis reported in the Emergency department file and the diagnosis reported at hospital discharge.
Length of hospital stay | Within hospital stay, maximum 21 days
Administration of non-invasive ventilation | Within hospital stay, maximum 21 days
Timing of non-invasive ventilation | Within hospital stay, maximum 21 days
Administration of diuretics | Within hospital stay, maximum 21 days
Timing of diuretics | Within hospital stay, maximum 21 days
Post emergency admission | Within hospital stay, maximum 21 days
  Type of department admitting the patient following emergency care (intensive care unit, cardiology unit, cardiac intensive care unit, post-emergency department, other...)
All-cause hospital mortality | Within hospital stay, maximum 30 days
Readmissions (all-cause and related to acute dyspnea) to the emergency department | Within 5 years after admission
Congestion score | Within 2 days of admission
  Assessed by: Congestion score assessed on chest X-ray on admission to the emergency department. The congestion score ranges from 0 (indicating no congestion signs) to 3 (indicating intense congestion).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU, Nancy, France